CLINICAL TRIAL: NCT06329531
Title: Validation of the Screen of Cancer Survivorship - Occupational Therapy Services (SOCS-OTS) Tool for Use in a Physical Medicine Rehabilitation Clinic
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0992; NCI-2024-02555 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Occupational Therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screen of Cancer Survivorship - Occupational Therapy Services (SOCS-OTS): You will be asked to complete three questionnaires and a short interview about yourself and how well you are able to complete your daily tasks. The SOCS-OTS, which is a 20-item questionnaire.
  Interventions: Other: Screen of Cancer Survivorship - Occupational Therapy Services (SOCS-OTS)

INTERVENTIONS:
Other: Screen of Cancer Survivorship - Occupational Therapy Services (SOCS-OTS) — Given by Questionnaire

SUMMARY:
To compare the results of the SOCS-OTS to another standardized screening measure that is currently being used by rehabilitation services at MD Anderson Cancer Center and to ensure that the SOCS-OTS correctly identifies those individuals needing OT services in cancer care.

DETAILED DESCRIPTION:
Primary Aim

1. Explore the SOCS-OTS for use in the Physical Medicine and Rehabilitation (PM&R) clinic by means of diagnostic testing including sensitivity and specificity.

Secondary Aims

1. Explore whether the SOCS-OTS identifies the likelihood that the presence or absence of OT referral is correctly predicted. To accomplish this, the likelihood ratios, and predictive values of the SOCS-OTS will be assessed.
2. Determine associations between the need for OT and demographic factors such as stage of cancer, cancer treatment etc.
3. Establish test-retest reliability of the SOCS-OTS.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 years an older
2. Currently medically followed in the PMR clinic (with or without acute disease)
3. Must speak and read English. The AM-PAC is currently validated in adults only. Additionally, the assessment tools are in English without translation into other languages, therefore only clients who do speak and read English will be included. Pregnant participants are not excluded.

Exclusion Criteria:

1. Potential participants with confusion and cognitive impairments that might hinder their ability to sign an informed consent form or participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer Participants
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Ekta Gupta, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org